CLINICAL TRIAL: NCT03448770
Title: To Compare Efficacy and Safety of Lactulose Versus Polyethylene Glycol for Treatment of Overt Hepatic Encephalopathy in Cirrhotics: A Randomized Controlled Trial
Brief Title: To Compare Efficacy and Safety of Lactulose Versus Polyethylene Glycol for Treatment of Overt Hepatic Encephalopathy in Cirrhotics.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-cirrhosis-14
Record Dates: First submitted 2018-02-19; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactulsoe (Active Comparator): Lactulose : 20-30gm 2-3 doses per day
  Interventions: Drug: Lactulose : 20-30gm
- Polyethlene Glycol (Experimental): PEG (Polyethlene Glycol)- 17 gm sachet 3-4 times per day
  Interventions: Drug: PEG- 17 gm sachet

INTERVENTIONS:
Drug: PEG- 17 gm sachet — PEG- 17 gm sachet 3-4 times per day
  Arms: Polyethlene Glycol
Drug: Lactulose : 20-30gm — Lactulose : 20-30gm
  Arms: Lactulsoe

SUMMARY:
All patients presenting to the emergency department of Institute of Liver and Biliary Sciences with known cirrhosis and hepatic encephalopathy with grade II will be included in the study. The patient will be randomized into one of the two arms of lactulose or polyethylene glycol. The patient on the lactulose arm will be administered 20 to 30 g of lactulose orally or by nasogastric tube (3 or more doses within 24 hours ) or if oral intake was not possible or inadequate. The Dose will be repeated to ensure 3-4 loose motions per day. The Polyethylene Glycol group will get 17 gm of PEG (Polyethylene Glycol) administered orally or via nasogastric tube. PEG (Polyethylene Glycol)will be administered in 3-4 doses in 24 hours to ensure 3-4 loose stools per day.

ELIGIBILITY:
Inclusion Criteria:

1. Documented cirrhosis with any underlying etiology
2. Hepatic encephalopathy of grade II and above
3. 18 to 65 years of age

Exclusion Criteria:

1. Acute change in mental status due to a diagnosis other than hepatic encephalopathy
2. Patients who have received lactulose as an anticoma measure before enrollment
3. Patient who have developed encephalopathy post bleed
4. Patients with gut paralysis
5. Patients with tense ascites
6. Patients with altered sensorium due to organic brain disease.
7. Patients with coexistent psychiatric illness that may hamper the proper assessment of hepatic encephalopathy
8. Hemodynamic instability obviating vasopressors for resuscitation
9. Acute liver failure defined as severe acute liver injury with encephalopathy and international normalized ratio (INR)≥1.5 in a patient without pre-existing liver disease
10. Refusal of consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Complete reversal of hepatic encephalopathy in both groups. | 3 days
  Complete reversal is defined as Grade 0 Encephalopathy

SECONDARY OUTCOMES:
Improvement in hepatic encephalopathy by two grades in both groups | 3 days
Length of Intensive Care Unit stay in both groups | 28 days
Adverse events in both groups | 3 days
Presence of encephalopathy changes in Electroencephalography in both groups | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided